CLINICAL TRIAL: NCT00388830
Title: "Emergency Bedside Ultrasonography of the Gallbladder: Does Fasting Matter?"
Brief Title: Emergency Ultrasound of the Gallbladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 26046
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Gallbladder Diseases
Keywords: Gallbladder; Ultrasound; Emergency Medicine
MeSH Terms: conditions — Gallbladder Diseases | interventions — High-Energy Shock Waves

INTERVENTIONS:
Procedure: Ultrasound

SUMMARY:
The purpose of this study is to determine whether fasting for 8 hours prior to ultrasonography for cholelithiasis (gallbladder pain) is needed.

DETAILED DESCRIPTION:
Ultrasonography of the gallbladder is currently the diagnostic modality of choice in determining cholelithiasis and cholecystitis. Historically this test has been performed in the Radiology suites where the patient was expected to fast for times of six to ten hours. Patients presenting to emergency departments (ED) have also been required to wait to have their study performed in order to have better visualization of the gallbladder. However, few studies have examined whether a fasting time matters in determining gallbladder pathology. Furthermore, with the emphasis on through-times in the ED, most EDs cannot afford holding their patients in the ED to wait for a test. Finally, with the advent of emergency bedside ultrasonography and the greater level of comfort emergency physicians (EP) have in diagnosing gallbladder pathology, it is possible to now determine an answer within minutes. We will test to see if EPs trained in the use of emergency bedside ultrasound can effectively and efficiently determine gallbladder pathology and if fasting has an impact on their ability to perform a quality ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 75
* Ability to consent for study

Exclusion Criteria:

* Inability to give informed consent
* Known pregnancy
* Prior cholecystectomy
* Inability to consume a fast food breakfast
* Known history of cholelithiasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
time to perform scan
diagnosis of pathology
performance of adequate measurement
overall adequacy of the scan

CONTACTS AND LOCATIONS:
Overall Officials: Robert O'Connor, MD, MPH, Study Director — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States